CLINICAL TRIAL: NCT00198666
Title: Efficacy of Zinc in the Treatment of Pneumonia in Hospitalized Children Less Than 2 Years of Age
Brief Title: Efficacy of Zinc in the Treatment of Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Mathuram Santosham, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H.22.03.01.06.A2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Pneumonia
Keywords: Pneumonia; zinc
MeSH Terms: conditions — Pneumonia | interventions — Zinc

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Children with severe pneumonia were randomly assigned to receive supplementation with elemental zinc.
  Interventions: Drug: Zinc
- Control (No Intervention): Children with severe pneumonia were randomly assigned to receive supplementation with placebo tablets.

INTERVENTIONS:
Drug: Zinc — Elemental Zinc
  Arms: Treatment

SUMMARY:
This study is designed to evaluate the efficacy of zinc supplementation in the treatment of children under the age of two years who have been hospitalized with severe pneumonia.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled clinical trial conducted between September 2003 and August 2004 at the Christian Medical College (CMC) Hospital in Vellore, India. CMC Hospital is a large teaching hospital and medical center that is accessed directly by the population of Vellore and adjoining districts and by referrals from local medical practitioners.

ELIGIBILITY:
Inclusion Criteria:

* children under two years old hospitalized with Pneumonia

Exclusion Criteria:

* healthy children

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 299 (Actual)
Dates: Start 2003-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Duration of severe symptoms | 2 years

SECONDARY OUTCOMES:
Time to recovery from severe pneumonia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mathuram Santosham, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

REFERENCES:
- [Derived] Coles CL, Bose A, Moses PD, Mathew L, Agarwal I, Mammen T, Santosham M. Infectious etiology modifies the treatment effect of zinc in severe pneumonia. Am J Clin Nutr. 2007 Aug;86(2):397-403. doi: 10.1093/ajcn/86.2.397. PMID 17684211